CLINICAL TRIAL: NCT04657107
Title: The Efficacy and Safety of S-ketamine in Elective Cesarean Section: a Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Study
Brief Title: The Efficacy and Safety of S-ketamine in Elective Cesarean Section
Acronym: ES-CS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Obstetrics and Gynecology Hospital (Other)
Collaborators: China Health Promotion Foundation (Unknown); Beijing Haidian Maternal and Child Health Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); The Fourth Hospital of Shijiazhuang (Other); Changzhi Maternal and Child Health Hospital (Unknown); Linfen Maternity&Child Healthcare Hospital (Unknown); Maternal and Child Health Hospital, Jiading District (Other); Tongzhou Maternal and Child Healthcare Hospital of Beijing (Unknown); Beijing Chaoyang District Maternal and Child Health Care Hospital (Unknown)
Responsible Party: Principal Investigator, Mingjun Xu, Chief of Anesthesiology department, Beijing Obstetrics and Gynecology Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BeijingOGH
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Anesthesia; Analgesia; Depression; Cesarean Section; Parturition
Keywords: S-ketamine; efficacy; safety; Postpartum depression
MeSH Terms: conditions — Agnosia; Depression; Depression, Postpartum | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Saline group (Placebo Comparator): Parturients were subsequently placed in a supine position with a left lateral tilt (15 ̊). Combined spinal-epidural anesthesia method (CSE) was performed at the L2-L3 or L3-L4 lumbar vertebral interspace, with 10～13mg 0.5% ropivacaine by a needle-through-needle technique. When adequate anesthesia to the T6 dermatome was achieved (Sensory and motor assessments were performed at 1 min intervals using pinprick testing and the modified Bromage score). Parturients received 10ml intravenous normal saline before surgery, If the anesthesia is inadequate, another 5ml 0.5% ropivacaine was given. Morphine hydrochloride 1 mg in saline 10 mL was injected by several times into the epidural space at the end of the operation. After the surgery, their PCA protocol consisted of 150 ug sufentanil and 24ml atropisetron diluted into 150 ml (2ml of basal infusion, a bolus of 0.5ml on demand, "lock-out" interval of 10 min, last for 48 h postoperatively);
  Interventions: Other: normal saline
- K1 group (Experimental): Parturients were subsequently placed in a supine position with a left lateral tilt (15 ̊). Combined spinal-epidural anesthesia method (CSE) was performed at the L2-L3 or L3-L4 lumbar vertebral interspace, with 10～13mg 0.5% ropivacaine by a needle-through-needle technique. When adequate anesthesia to the T6 dermatome was achieved (Sensory and motor assessments were performed at 1 min intervals using pinprick testing and the modified Bromage score). Parturients received 10ml intravenous 0.2mg/kg before surgery, If the anesthesia is inadequate, another 5ml 0.5% ropivacaine was given. Morphine hydrochloride 1 mg in saline 10 mL was injected by several times into the epidural space at the end of the operation. After the surgery, their PCA protocol consisted of 150 ug sufentanil and 24ml atropisetron diluted into 150 ml (2ml of basal infusion, a bolus of 0.5ml on demand, "lock-out" interval of 10 min, last for 48 h postoperatively);
  Interventions: Drug: S-ketamine
- K2 group (Experimental): Parturients were subsequently placed in a supine position with a left lateral tilt (15 ̊). Combined spinal-epidural anesthesia method (CSE) was performed at the L2-L3 or L3-L4 lumbar vertebral interspace, with 10～13mg 0.5% ropivacaine by a needle-through-needle technique. When adequate anesthesia to the T6 dermatome was achieved (Sensory and motor assessments were performed at 1 min intervals using pinprick testing and the modified Bromage score). Parturients received 10ml intravenous 0.3mg/kg before surgery, If the anesthesia is inadequate, another 5ml 0.5% ropivacaine was given. Morphine hydrochloride 1 mg in saline 10 mL was injected by several times into the epidural space at the end of the operation. After the surgery, their PCA protocol consisted of 150 ug sufentanil and 24ml atropisetron diluted into 150 ml (2ml of basal infusion, a bolus of 0.5ml on demand, "lock-out" interval of 10 min, last for 48 h postoperatively);
  Interventions: Drug: S-ketamine

INTERVENTIONS:
Drug: S-ketamine — K1 group: pregnant women received 0.2mg/kg S-ketamine, intravenous drip;
  Other Names: esketamine
  Arms: K1 group
Other: normal saline — Saline group: pregnant women received saline, intravenous drip
  Other Names: physiological saline
  Arms: Saline group
Drug: S-ketamine — K2 group: pregnant women received 0.3mg/kg S-ketamine, intravenous drip;
  Other Names: esketamine
  Arms: K2 group

SUMMARY:
During the past years, a large number of clinical trials have investigated the use of the non-competitive N-methyl-D-aspartate (NMDA) receptor antagonist racemic ketamine as an adjunct to local anaesthetics, opioids, or other analgesic agents for the management and prevention of postoperative pain. Actually racemic ketamine not only abolishes peripheral afferent noxious stimulation, but can also prevent the central nociceptor sensitization. S-ketamine, one of two enantiomers of racemic ketamine, has twice the analgesic potency of the racemate. Moreover, S-ketamine shows smaller nervous system and less psychotropic effects than racemic ketamine , which may make the drug more suitable for clinical use. Recently, S-ketamine has been approved to treat refractory depression (TRD) and major depressive disorder (MDD) by the FDA .S-ketamine may have greater clinical significance due to the high rate of maternal depression. Therefore, we plan to explore whether clinical use of S-ketamine can optimize anesthesia protocol and improve maternal prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. ASA II;
2. Parturients voluntarily sign an informed consent form, fully understands the purpose and significance of the study, and voluntarily abides by the clinical study procedure;
3. Subjects who plan to be elected to undergo cesarean section under continuous combined spinal-epidural anesthesia;
4. Age 18 to 40 years;
5. The expected duration of surgery was less than 2h;
6. Prenatal body mass index (BMI) was less than 35kg/m2。

Exclusion Criteria:

1. Parturients with contraindications to continuous combined spinal-epidural anesthesia (such as history of central nervous system infection, spinal cord or spinal canal disease or surgery history, systemic infection, skin or soft tissue infection at the puncture site, coagulation dysfunction);
2. Those who have a history of stroke, cognitive dysfunction, and epilepsy;
3. Patients with a history of myocardial infarction, angina pectoris, or a serious arrhythmia such as second-degree and above-degree atrioventricular block within 6 months before screening;
4. Pregnancy with other diseases (malignant tumors, hypertension during pregnancy, abnormal thyroid function, etc.);
5. In the non-oxygen state, the peripheral blood oxygen saturation (SpO2) <92%;
6. Subjects whose prolactin is greater than the upper limit of normal during the screening period;
7. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), glutamine transferase (GGT)> 1.5 times than the normal value, and total bilirubin is higher than the upper limit of normal value, and blood creatinine (Cr)>1.2 times than the upper limit of normal value;
8. The effect of combined spinal-epidural anesthesia is not good, and other anesthetics are needed;
9. People with a history of allergies to various foods and drugs;
10. Continuous taking for any reason within 3 months before the screening, including but not limited to: ketamine, non-steroidal anti-inflammatory drugs (aspirin, acetaminophen, indomethacin, diclofenac, ibuprofen, parecoxib) Sodium, etc.), alpha adrenergic receptor agonists (dexmedetomidine hydrochloride, clonidine, etc.), glucocorticoids (dexamethasone hydrochloride, hydrocortisone, methylprednisolone, etc.), antiepileptic ( Carbamazepine, sodium valproate, etc.), sedation (diazepam, estazolam, midazolam, alprazolam, barbital, phenobarbital and chloral hydrate, etc.), Chinese herbal medicine or Chinese patent medicine with pain and sedative effect;
11. There is a history of drug abuse and/or alcohol abuse within 1 year before the screening;
12. Participated in other drug or device trials within 3 months before the screening;
13. Subjects judged by the investigator to be unsuitable to participate in this clinical study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Parturients undergoing elective cesarean section
Enrollment: 402 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative anesthesia effect | Day 1
  Anesthesia effect is graded I-IV. Level I means that it is very satisfactory, while Level IV means other anesthesia methods are needed to complete the operation. We expect to reach level I.
Ramsay Sedation Scale score | Day 1
  The Ramsay Sedation Scale (RSS) was the first scale to be defined for sedated patients and was designed as a test of rousability. The RSS scores sedation at six different levels, according to how rousable the patient is.
Clock-in-the-Box(CIB) | Day 0 & Day 2
  The Clock-in-the-Box (CIB) is a rapidly administered cognitive screening measure which has been previously validated with cognitive screening and neuropsychological assessments. The CIB is scored on a 0-8 point scale and the total score includes two separate subscale scores. The higher scores reflect better performance.

SECONDARY OUTCOMES:
PHQ-9 | Day 0 & Day 3 & Day 8 & Day 43
  PHQ-9 is the major depressive disorder(MDD) module of the full PHQ. Used to provisionally diagnose depression and grade severity of symptoms in general medical and mental health settings. Scores each of the 9 DSM criteria of MDD as "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score. Higher PHQ-9 scores are associated with decreased functional status and increased symptom-related difficulties, sick days, and healthcare utilization.
Edinburgh Postnatal Depression Scale(EPDS) | Day 3 & Day 8 & Day 43
  EPDS is a valuable and efficient way of identifying patients at risk for "perinatal" depression. Mothers who score above 13 are likely to be suffering from a depressive illness of varying severity depression.
Apgar score | Day 0
  The Apgar score is a test given to newborns soon after birth. This test checks a baby's heart rate, muscle tone, and other signs to see if extra medical care or emergency care is needed. The test is usually given twice: once at 1 minute after birth, and again at 5 minutes after birth.
placental transfer of S-ketamine | Day 0
  Placental transfer was evaluated based on the whole blood concentrations of S-ketamine in the maternal and cord blood
blood gas | Day 0
  Blood gases are a group of tests that are performed together to measure the pH and the amount of oxygen (O2) and carbon dioxide (CO2) present in a sample of blood
umbilical arterial (UA)/umbilical venous (UV) ratio | Day 0
  UA/UV ratio was evaluated based on the blood concentrations of S-ketamine in the umbilical arterial and umbilical venous blood

CONTACTS AND LOCATIONS:
Overall Officials: Lei Wang, Principal Investigator — Beijing Haidian Maternal and Child Health Hospital; Shaoqiang Huang, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University; Jin Zhang, Principal Investigator — The Fourth Hospital of Shijiazhuang; Yingbin Ren, Principal Investigator — Changzhi Maternal and Child Health Hospital; Yong Qin, Principal Investigator — Linfen Maternity&Child Healthcare Hospital; Shenghua Li, Principal Investigator — Maternal and Child Health Hospital, Jiading District; Zhenhuan Hou, Principal Investigator — Tongzhou Maternal and Child Healthcare Hospital of Beijing; Shuyi Miao, Principal Investigator — Beijing Chaoyang District Maternal and Child Health Care Hospital